CLINICAL TRIAL: NCT02214849
Title: LATCH: Lactation Advice Thru Texting Can Help
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1206010472
Record Dates: First submitted 2014-08-01; First posted 2014-08-12 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Breastfeeding Support
Keywords: Breastfeeding; Breastfeeding peer counseling; Exclusive breastfeeding; Formula supplementation; Mobile health; WIC program
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LATCH Intervention (Experimental): Women enrolled in the WIC program and receiving breastfeeding peer counseling services will receive text messages to support them with their breastfeeding intentions. They will start receiving automated text messages starting in pregnancy and continuing throughout the first 6 months after giving birth. Messaging during pregnancy will emphasize what to expect in the hospital, the onset of lactation, skin-to-skin contact with baby, early and often breastfeeding in post-partum period, milk transfer (suck & swallow), positioning (with links), common breastfeeding problems and how to seek help. Throughout the study, participants will be able to respond to automated text messages with specific questions that will be received and answered by their WIC program peer counselors. Texting will also have prompts to respond occasionally (at minimum once every two weeks) to ensure that phone is still in service and that the participant in the intervention arm are receiving intervention.
  Interventions: Behavioral: LATCH Intervention

INTERVENTIONS:
Behavioral: LATCH Intervention

SUMMARY:
The purpose of this study is to find out if a two-way texting platform to be used as an adjunct tool for breastfeeding peer counselors can improve breastfeeding behaviors among women enrolled in the WIC program in Connecticut. The hypothesis of the study is that providing additional information and support through text messaging starting in pregnancy and continuing after the birth of the child will increase exclusive breastfeeding rates during the first six months of life.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women > 18 years
* Prenatal intention to breastfeed
* Prenatal enrollment < 28 weeks gestation
* Have an unlimited text message cell phone plan
* Knows how to send a text message
* 5th grade literacy level

Exclusion Criteria:

* Lack of fluency in either English or Spanish
* Infant born premature (<37 weeks)
* > 3 days in NICU
* Any major maternal-newborn medical problem affecting breastfeeding
* Birth weight <5lbs

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 249 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Exclusive Breastfeeding Rate | 2 weeks after birth
Change in Exclusive Breastfeeding Rate | 3 months after birth
Change in Exclusive Breastfeeding Rate | 6 months after birth

SECONDARY OUTCOMES:
Chance in the Percent of WIC Participants Reached by Breastfeedng Counselor | 48 hours after giving birth
Change in Number of Contact Between WIC Participants and Breastfeeding Peer Counselors | 2 weeks after birth
Change in Number of Contact Between WIC Participants and Breastfeeding Peer Counselors | 3 months after birth
Change in Number of Contact Between WIC Participants and Breastfeeding Peer Counselors | 6 months after birth
Change in breastfeeding self-efficacy | 2 weeks after birth
  Self-efficacy refers to an individuals' confidence in their capability to initiate, maintain, and (if stopped) re-start breastfeeding. It will be measured with the scale proposed by Schwarzer. Self-efficacy scale includes 5 questions, each with 4 response options ranging from "very false" to "very true". Average score will be generated by summing responses to questions 1 through 5 and dividing by the total number of questions. Average scores will range from 1 to 4. The higher the score the better the level of self-efficacy.
  Reference: Schwarzer R. Modeling health behavior change: How to predict and modify the adoption and maintenance of health behaviors. Applied Psychology: An International Review. 2008 2008;57(1):1-29.
Change in breastfeeding self-efficacy | 3 months after birth
Change in breastfeeding self-efficacy | 6 months after birth
Change in breastfeeding action planning | 2 weeks
  Action planning refers to the "when", "where", and "how" of the behavior or the sequence of events making up breastfeeding behaviors. It will be measured with the scale proposed by Schwarzer. Action planning scale includes 7 questions, each with 4 response options ranging from "very false" to "very true". An average score will be generated by summing responses to questions 1 through 7 and dividing by the total number of questions. Average scores will range from 1 to 4. The higher the score the better the level of action planning.
  Reference: Schwarzer R. Modeling health behavior change: How to predict and modify the adoption and maintenance of health behaviors. Applied Psychology: An International Review. 2008 2008;57(1):1-29.
Change in breastfeeding action planning | 3 months
Change in breastfeeding action planning | 6 months
Change in breastfeeding coping planning | 2 weeks
  Coping planning refers to the identification of potential barriers to engaging in and maintaining breastfeeding behavior and the extent to which an individual has developed strategies to cope with those barriers. It will be measured with the scale proposed by Schwarzer. Coping planning scale includes 6 questions, each with 4 response options ranging from "very false" to "very true". An average score will be generated by summing responses to questions 1 through 6 and dividing by the total number of questions. Average scores will range from 1 to 4. The higher the score the better the level of coping planning.
  Reference: Schwarzer R. Modeling health behavior change: How to predict and modify the adoption and maintenance of health behaviors. Applied Psychology: An International Review. 2008 2008;57(1):1-29.
Change in breastfeeding coping planning | 3 months
Change in breastfeeding coping planning | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Perez-Escamilla, PhD, Principal Investigator — Yale University; Nurit Harari, MD, Study Director — Yale University
Locations (1):
- Yale School of Public Health, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276